CLINICAL TRIAL: NCT04499209
Title: A Phase 1, Single-Center, Randomized, Placebo-Controlled, Ascending Single-Dose Study of the Pharmacokinetics, Safety, and Tolerability of Oral XG005 in Healthy Volunteers
Brief Title: Pharmacokinetics Study of XG005 Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xgene Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: XG005-01
Record Dates: First submitted 2020-07-13; First posted 2020-08-05 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: Period 1: ascending single-dose of XG005 vs Placebo; Period 2: combination of Naproxen and Pregabalin
Who Masked: Participant, Investigator
Masking Description: Period 1: Participants and investigators were blinded Period 2: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Period 1- XG005 (Experimental): XG005 capsule in 4 dose level
  Interventions: Drug: XG005
- Period 2- Naproxen and Pregabalin (Active Comparator): Combination of Naproxen and Pregabalin
  Interventions: Drug: Combination of Naproxen and Pregabalin
- Period 1- Placebo (Placebo Comparator): XG005 matching placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: XG005 — XG005 Capsule
  Arms: Period 1- XG005
Drug: Combination of Naproxen and Pregabalin — Naproxen and Pregabalin are commercially available products with trade names of Aleve and Lyrica
  Arms: Period 2- Naproxen and Pregabalin
Drug: Placebos — Placebo Capsule
  Arms: Period 1- Placebo

SUMMARY:
This was a Phase 1, single-center, randomized, placebo-controlled, 2-period, ascending single-dose study assessing the PK, safety, and tolerability of single ascending doses of XG005 (Period 1) and the naproxen and pregabalin combination (Period 2), in 5 dose groups each with 10 subjects.

DETAILED DESCRIPTION:
Period 1 was double-blind and randomized 8 subjects (1:1 allocation ratio by gender) to XG005 and 2 subjects (1:1 allocation ratio by gender) to placebo. Subjects were enrolled sequentially into a total of 5 ascending dose levels pending safety review, and PK review where possible, of Period 1 of the prior dose level. Sentinel dose participants (1 for XG005 and 1 for placebo) were included as the first dose administered at each dose level in Period 1.

In Period 2, all subjects in the last three XG005 dose groups received approximate molar equivalents of naproxen and pregabalin corresponding to XG005 doses after a 7-day washout period. Period 2 was open-label with 10 subjects per group.

PK blood samples in each treatment period were collected at 0 (pre-dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hrs after drug administration.

ELIGIBILITY:
Inclusion Criteria:

* BMI range of 18-30 kg/m2
* Medically healthy subjects
* Creatinine clearance ≥ 80 mL/min

Exclusion Criteria:

* History or presence of significant diseases
* History or presence of alcoholism or drug abuse
* Consumption of alcohol 48 hours prior each dose
* Hypersensitivity or idiosyncratic reaction to the study drug
* Abnormal diet (for whatever reason) during the 30 days prior to the first dosing;
* Donation (standard donation amount or more) of blood or blood products
* Plasma donation within 7 days prior to the study;
* Participation in another clinical trial within 30 days prior to the first dose;
* Female subjects who are pregnant or lactating;
* Hemoglobin < 120 g/L

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | Day1 to Day 4
Time to maximum concentration (Tmax) | Day1 to Day 4
Area under the concentration-time curve from time 0 to last measurable time-point (AUC0-t) | Day1 to Day 4
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | Day1 to Day 4
Terminal Elimination Rate Constant (kel) | Day1 to Day 4
Terminal half-life (t1/2) | Day1 to Day 4
Terminal clearance (CL/F) | Day1 to Day 4
Volume of distribution (Vd/F) | Day1 to Day 4

SECONDARY OUTCOMES:
incidence and severity of adverse events (AEs) | Day -1 to Day 8
blood pressure | Day -1 to Day 8
  vital signs
heart rate | Day -1 to Day 8
  vital signs
respiratory rate | Day -1 to Day 8
  vital signs
temperature | Day -1 to Day 8
  vital signs
physical examination | Day -1 to Day 8
  Cardiovascular, Ears, Nose and Throat, Eyes, Gastrointestinal, Head, Lymph Nodes, Musculoskeletal, Neurological, Respiratory, Skin
electrocardiogram (ECG) parameters; | Day -1 to Day 8
  ECG-PR, RR, QRS, QT, and QTc intervals
clinical laboratory parameters -chemistry | Day -1 to Day 8
  BUN, Creatinine, Total bilirubin, Total protein, Alkaline phosphatase, Uric Acid, Estimated creatinine clearance, Creatine Phosphokinase (CPK), AST (SGOT), ALT (SGPT), Glucose, Sodium, Potassium
clinical laboratory parameters- hematology | Day -1 to Day 8
  Hemoglobin, Hematocrit, Red Blood Cell Count, White Blood Cell Count with differential, Platelet Count
clinical laboratory parameters urinalysis | Day -1 to Day 8
  * pH • Specific gravity • Protein
  * Glucose • Ketones • Bilirubin
  * Blood • Nitrite • Urobilinogen
  * Leukocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research Ltd, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No